CLINICAL TRIAL: NCT04716816
Title: Pain Relief Following Stripping Massage for Rhomboid Myofascial Trigger Points After Thoracoscopic Surgery
Brief Title: Stripping Massage After Thoracoscopy
Acronym: SMAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202011061RINA
Record Dates: First submitted 2021-01-17; First posted 2021-01-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Chest Pain
Keywords: Chest pain; Stripping massage; thoracoscopy; trigger points
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: treatment method and treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional treatment (No Intervention): received conventional analgesics.
- Stripping massage (Experimental): received SM twice daily in the active trigger points of the rhomboid for two weeks.
  Interventions: Procedure: Stripping massage

INTERVENTIONS:
Procedure: Stripping massage — Stripping massage for rhomboid myofascial trigger points
  Arms: Stripping massage

SUMMARY:
This study investigated the effects of stripping massage (SM) on myofascial trigger points in the rhomboid after thoracoscopic surgery.

DETAILED DESCRIPTION:
This study investigated the effects of stripping massage (SM) on myofascial trigger points in the rhomboid after thoracoscopic surgery. Sixty patients with chest pain after thoracoscopic surgery were randomized divided into two equal groups (A and B). Group A (n = 100) received conventional analgesics. Group B (n = 100) received SM twice daily in the active trigger points of the rhomboid for two weeks. The visual analogue scale, a pressure algometer, will be used to evaluate patients' pre- and post-treatment statuses.

This study will compare differences between the current traditional method (using analgesics) and the SM for rhomboid myofascial trigger points for post-thoracoscopic chest pain, and analyze the variables generated by the two different methods including demand time of analgesics, acceptance, and differences of visual analogue scale. The results of the study will use scientific data to prove which way is a good way to take into account of the relief of patient's chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain with visual analogue scale larger than 3 after thoracoscopic surgery

Exclusion Criteria:

* bleeding tendency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-17 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores on the Visual Analog Scale | baseline, 3 days, one weeks, two weeks, one month
  differences of visual analogue scale. (score from mild 0 to severe 10)

SECONDARY OUTCOMES:
demand time of analgesics | baseline, 3 days, one weeks, two weeks, one month
  demand time of analgesics after thoracoscopic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Ming Huang, MD, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Research Ethics Committee, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No